CLINICAL TRIAL: NCT06587763
Title: Late Biomarkers in Adult Survivors After Out-of-hospital Cardiac Arrest
Status: Not yet recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); University of Helsinki (Other)
Responsible Party: Sponsor
Other Study IDs: STEPCARE late biomarker study
Record Dates: First submitted 2024-06-18; First posted 2024-09-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Biomarkers; Brain injury; Inflammation; Dementia
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Brain Injuries; Inflammation; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and PAX-RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood samples are collected at six months follow-up from adult survivors after out-of-hospital cardiac arrest. Patients will be informed about the study and if they consent to participation, venous blood will be drawn by authorised medical personnel. Plasma, serum and PAX-RNA will be collected (ca 15 ml in total), processed and frozen for analysis after trial completion.

DETAILED DESCRIPTION:
Blood samples are collected at six months follow-up from adult survivors after out-of-hospital cardiac arrest. Patients will be informed about the study and if they consent to participation, venous blood will be drawn by authorised medical personnel. Plasma, serum and PAX-RNA will be collected (ca 15 ml in total), processed and frozen for analysis after trial completion.

Samples will be analysed in batch for biomarkers of brain injury, inflammation etc.

Primary outcome is functional outcome (modified Rankin Scale 4-6) at six months after cardiac arrest.

Secondary outcomes are neurocognitive function according to the Montreal Cognitive Assessment (MoCA), Symbol Digits Modalities Test (SDMT).

ELIGIBILITY:
Inclusion Criteria:

* Survivors of out-of-cardiac arrest who participate in the extended follow-up study of the STEPCARE trial at selected sites only

Exclusion Criteria:

* Patients not participating in the extended follow-up at participating sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an out-of-hospital cardiac arrest who survived to six months follow-up
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 6 months
  Modified Rankin Scale 4-6

SECONDARY OUTCOMES:
Neurocognitive outcomes | 6 months
  Montreal Cognitive Assessment
Neurocognitive outcomes | 6 months
  Symbol Digit Modalities Test

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Helsingborgs Hospital, Helsingborg
  - Skåne university hospital, Lund
  - Skåne University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request after publication of results.

REFERENCES:
- See also: trial Homepage — http://www.stepcare.org